CLINICAL TRIAL: NCT03639844
Title: Expanded Access Protocol for CaspaCIDe T Cells From An HLA-Partially Matched Related Donor After Negative Selection of TCR αβ+T Cells In Pediatric Patients Affected by Hematological and Other Disorders
Brief Title: BPX-501 T Cells Infused Post Stem Cell Transplant in Pediatrics With Non-Malignant Disorders Ineligible for BPU004 Study
Status: No longer available | Type: Expanded Access
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: BP-C-004
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Hurler Syndrome; Inherited Metabolic Disorder; Lysosomal Storage Disorder; Metachromatic Leukodystrophy; Inborn Errors of Metabolism
MeSH Terms: conditions — Mucopolysaccharidosis I; Lysosomal Storage Diseases; Leukodystrophy, Metachromatic; Metabolism, Inborn Errors | interventions — AP 1903 reagent; Injections

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: rivogenlecleucel — BPX-501 T cells are genetically modified with a suicide safety switch. The cells are infused after T cell-depleted HSCT to potentially enhance immune reconstitution while reducing severity and duration of GVHD.
  Other Names: BPX-501 T cells
Drug: rimiducid — Rimiducid induces activation of the Caspase 9 suicide gene in BPX-501 T cells inducing apoptosis of the modified T cells in case of GVHD
  Other Names: AP1903; Rimiducid for Injection; AP1903 for Injection

SUMMARY:
Providing access of BPX-501 gene modified T cells and rimiducid to pediatric patients who do not meet the eligibility criteria of the BP-U-004 study.

DETAILED DESCRIPTION:
This is an expanded access protocol of BPX-501 T cells infused after T cell-depleted HSCT in pediatric patients with non-malignant hematologic disorders eligible for treatment on the BP-U-004 study.

The purpose of this protocol is to provide access to the CaspaCIDe system combination product (BPX-501 gene modified T cells and rimiducid) to patients on a case by case basis who do not meet the BP-U-004 protocol eligibility criteria. BPX-501 infusion can enhance immune reconstitution with the potential for reducing the severity and duration of severe acute GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females
2. Age < 21 years and > 3 months
3. Life expectancy > 10 weeks
4. Patients deemed eligible for allogeneic stem cell transplantation.
5. Non-malignant disorders including:

   1. inherited metabolic disorders such as adrenal leukodystrophy;
   2. lysosomal storage disorders such as Hurler syndrome or metachromatic leukodystrophy
   3. other inborn errors of metabolism
6. Lack of suitable conventional donor (HLA identical sibling or HLA phenotypically identical relative evaluated using high resolution molecular typing).
7. A minimum genotypic identical match of 5/10 is required.
8. The donor and recipient must be identical, as determined by high resolution typing, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, and HLA- DRB1.
9. Lansky/Karnofsky score > 50
10. Signed written informed consent

3.2 Subject exclusion criteria

1. Age < 3 months or >21 years
2. Patients with non-malignant disorders eligible for treatment on the BP-U-004 study:

   1. primary immune deficiencies,
   2. severe aplastic anemia not responding to immune suppressive therapy,
   3. osteopetrosis,
   4. selected cases of hemoglobinopathies and
   5. congenital/hereditary cytopenia, including Fanconi Anemia before any clonal malignant evolution (MDS, AML)
3. Greater than Grade II acute GVHD or chronic extensive GVHD due to a previous allograft at the time of inclusion
4. Patient receiving an immunosuppressive treatment for GVHD treatment due to a previous allograft at the time of inclusion
5. Dysfunction of liver (ALT/AST > 5 times normal value, or bilirubin > 3 times normal value), or of renal function (creatinine clearance < 30 ml / min)
6. Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or left ventricular ejection fraction < 40%)
7. Current active infectious disease (including positive HIV serology or viral RNA)
8. Serious concurrent uncontrolled medical disorder
9. Pregnant or breast feeding female patient
10. Lack of parents'/guardian's informed consent.

    -

Ages: 3 Months to 21 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals, Study Director — Bellicum Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University; Division of Pediatric Stem Cell Transplant & Regenerative Medicine, Palo Alto, California